CLINICAL TRIAL: NCT01105468
Title: Leistungsbewertungsprüfung: Atemluftanalyse für Die Diagnose Von Brustkrebs, für Die Überwachung Der Therapie Und für Die Voraussage Des Metastasenrisikos
Brief Title: Breath Gas Analysis for the Diagnosis of Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: Sponsor quit partnership in Oncotyrol-Center for Personalized Medicine, and consequential loss of public funding.
Sponsor: Ionimed Analytik GmbH (Industry)
Collaborators: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: BC1
Record Dates: First submitted 2010-04-08; First posted 2010-04-16 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Mamma Carcinoma
Keywords: Breath gas analysis; Volatile components in exhaled breath

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Mamma Carcinoma, no treatment
  Interventions: Device: Breath Collecting Unit
- Mamma Carcinoma, treatment
  Interventions: Device: Breath Collecting Unit
- No Mamma Carcinoma diagnosed by X-ray
  Interventions: Device: Breath Collecting Unit

INTERVENTIONS:
Device: Breath Collecting Unit — Collect two breath gas samples per patient on one day before surgery
  Other Names: BCU
  Groups: Mamma Carcinoma, no treatment; No Mamma Carcinoma diagnosed by X-ray
Device: Breath Collecting Unit — Collect two or more breath gas samples on different days during adjuvant or neo-adjuvant therapy.
  Other Names: BCU
  Groups: Mamma Carcinoma, treatment

SUMMARY:
The volatile content of the exhaled breath gas of mamma carcinoma patients will be chemically analyzed by proton-transfer-reaction time of flight mass spectrometry.

The goal of the study is to determine typical breath gas components that allow to distinguish patients with mamma carcinoma from women without carcinoma. Further, the investigators will test whether these breath gas markers can be used as tumor markers, which change in a typical manner during the progress of the disease. Finally the data will be investigated for the presence of marker components, that identify patients who will develop metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Mamma carcinoma diagnosed by histology (cases)
* Mamma carcinoma excluded by radiology (controls)
* At the time of diagnosis before surgery
* At the beginning and during chemotherapy;

Exclusion Criteria:

* No informed consent form singed

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2010-04; Primary Completion 2013-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Breath gas markers | 3 years
  Breath gas markers that allow to distinguish patients with mamma carcinoma from women without carcinoma;

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gynecology and Obstetrics, Medical University Innsbruck, Innsbruck, Tyrol, Austria